CLINICAL TRIAL: NCT02637310
Title: A Multi Center, Randomized, Double-blind, Placebo-controlled, Parallel, Phase 2b Clinical Trial to Evaluate the Efficacy and Safety of N02RS1 in Patients With Acute Bronchitis
Brief Title: Evaluate the Efficacy and Safety of N02RS1 in Patient With Acute Bronchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMK-N02RS1_Phase 2B
Record Dates: First submitted 2015-12-08; First posted 2015-12-22 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N02RS1 1200mg (Experimental): Combination of Broussonetia spp and Lonicera spp
  Interventions: Drug: N02RS1 1200mg
- Placebo (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N02RS1 1200mg — 1200mg/day, Three times a day orally, 2 tablets once, 7 days
  Arms: N02RS1 1200mg
Drug: Placebo — 1200mg/day, Three times a day orally, 2 tablets once, 7 days
  Arms: Placebo

SUMMARY:
A multi center, randomized, double-blind, placebo-controlled, parallel, phase 2b clinical trial to evaluate the efficacy and safety of N02RS1 in patients with acute bronchitis

DETAILED DESCRIPTION:
Suitable subjects randomized to the experimental or control group. The subjects eat IP during 7days. Visit 3(3 days) evaluate BSS through phone call and visit 4(8 days) evaluate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19, under 75 of age
* Patients acute bronchitis, sputum symptoms, BSS over 7 points.
* Patients acute bronchitis within 7days.
* Non-pregnant, patients who agree to contraception.
* Patients who can write diary and available to communicate.
* Patients voluntarily agreed

Exclusion Criteria:

* Patients with hypersensitivity to the drug.
* Patients who have gotten systemic steroid treatment within 4 weeks.
* Patients who have gotten treatment of antibiotics, bronchodilators, painkiller and secretagog within 7 days.
* Patients who have gotten treatment of mucus solvents or antitussives within 3 days.
* Patients who serious respiratory infections requiring antibiotic treatment, allergic bronchial asthma, bronchiectasis and chronic obstructive pulmonary disease.
* Patients heart disease, severe kidney, liver disease.
* The bleeding tendency or immunosuppressed patients.
* Patients with clinically significant abnormal values.
* Pregnant women or nursing mothers.
* Patients alcoholics or drug abuse.
* Patients taking other clinical trail's medicines within 30 days.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
BSS(Bronchitis Severity Score) score variation compared to baseline after 7 days | Visit 1(-3days, screening), 2(0day, randomization), 3(3days), 4(8days)